CLINICAL TRIAL: NCT01326117
Title: Daily Tadalafil and Gastric Emptying Time in Diabetic Gastroparesis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of patients who meet inclusion criteria; there was one screen failure
Sponsor: Mark Feinglos (Other)
Collaborators: Duke University (Other); Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Mark Feinglos, Division Chief, Department of Endocrinology, Diabetes, and Metabolism, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00027389
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Gastroparesis; Diabetic Gastroparesis; Nausea; Vomiting
Keywords: gastroparesis; gastric emptying; diabetes; Stomach Diseases; Gastrointestinal Diseases; Digestive System Diseases; Phosphodiesterase Inhibitors; Neurologic Manifestations; Paralysis; Signs and Symptoms; Pharmacologic Actions
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting; Diabetes Mellitus; Stomach Diseases; Gastrointestinal Diseases; Digestive System Diseases; Neurologic Manifestations; Paralysis; Signs and Symptoms | interventions — Tadalafil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- tadalafil (Experimental)
  Interventions: Drug: tadalafil

INTERVENTIONS:
Drug: tadalafil — 7 days of Cialis for Daily Use (5mg)
  Other Names: Cialis

SUMMARY:
The investigators hypothesize that in adult patients with diabetic gastroparesis with Type 1 diabetes (HbA1c ≤ 10.5%), daily tadalafil use will significantly improve gastric emptying compared to baseline as measured by gastric emptying time.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosis
* Age 18 - 65 years (inclusive)
* Hemoglobin A1c ≤ 10.5% within the last 4 months
* Diagnosis of gastroparesis, or symptoms consistent with gastroparesis (early satiety, chronic intermittent nausea or vomiting with food intake)
* Patient has gastroparesis confirmed on screening study
* A female patient is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea, or child-bearing potential with negative serum hCG prior to each gastric emptying study.

Exclusion Criteria:

* Active nitrate use (e.g. Cialis, Viagra, Levitra, nitroglycerin, Isordil, Imdur, amyl nitrate/poppers)
* Fasting fingerstick glucose > 250 mg/dL
* History of abdominal surgery including gastric banding procedure
* Patient is on chronic parenteral feeding
* Patient has a history of eating disorders (anorexia nervosa, binge eating, bulimia)
* Regular opiate use
* Recent (last 6 weeks) history of poor control of diabetes e.g. hypoglycemia requiring medical intervention, diabetic ketoacidosis, admission for control diabetes or complications of diabetes
* Acute severe gastroenteritis
* The patient has participated in another clinical trial in the last 30 days.
* Use of medications potentially influencing upper gastrointestinal motility or appetite within one week of the study [e.g., prokinetic drugs, macrolide antibiotics (erythromycin), GLP-1 mimetics/analog, amylin analog]
* History or presence of clinically significant gastro-intestinal, hepatic or renal disease or other condition that would in the opinion of the investigator make the subject unsuitable for inclusion in this clinical study.
* Chronic angina or NYHA class III or IV CHF
* Concurrent use of ketoconazole or itraconazole
* History of severe vision loss, retinitis pigmentosa, or non-arteritic anterior ischemic optic neuropathy (NAION)
* History of CVA
* Pregnant females as determined by positive serum hCG test
* Lactating females
* Uncontrolled hypertension (SBP > 160 or DBP > 100)
* Hypotension (SBP < 90 or DBP < 60)
* Other major medical conditions: priapism, sickle cell anemia, multiple myeloma, leukemia, active cancer diagnosis, HIV/AIDS, alcoholism, or bleeding diathesis.
* Intolerance to active or inactive ingredients of Cialis, or intolerance to other PDE-5 inhibitors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
improvement in Gastric Emptying Study residual tracer amount | 7 days with intervention
  change in gastric emptying compared to baseline as measured by gastric emptying time.

CONTACTS AND LOCATIONS:
Overall Officials: Mark N Feinglos, MD, CM, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States